CLINICAL TRIAL: NCT00417768
Title: Safety and Effectiveness of Local Instillation of tPA in the Management of Complex Intra-abdominal Fluid Collections: a Randomized, Double Blinded Controlled Clinical Trial
Brief Title: Safety and Effectiveness of tPA in Intra-abdominal Abscesses
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Change in patient population no longer fit study criteria.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-0238-E
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Abscess
Keywords: tissue plasminogen activator; intraabdominal; abscess; percutaneous drainage
MeSH Terms: conditions — Abscess | interventions — Tissue Plasminogen Activator; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tissue Plasminogen Activator (Active Comparator): tPA administered by drainage tube into abscess, allowed to dwell for one hour and then drained into drainage bag. Dose of tPA administered to be determined by the volume of drainage immediately post drain insertion. This intervention is done on day 0, 1 and 2.
  Interventions: Drug: Tissue Plasminogen Activator
- Instillation of Normal Saline (Sham Comparator): Insertion of abdominal drainage tube to drain intra-abdominal abscess. Normal Saline administered immediately post drain insertion. Normal Saline (10 cc) allowed to dwell for one hour, then allowed to drain into drainage bag.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Tissue Plasminogen Activator — The dosage of tPA is determined by the volume of drainage obtained when abscess is first drained. The same dose will be repeated on day 1 and 2.
  Other Names: Intra-abdominal drainage; tPA
  Arms: Tissue Plasminogen Activator
Other: Normal Saline — Normal Saline will be used rather than Tissue Plasminogen Activator for the Sham arm.
  Other Names: Intra-abdominal abscess drain; sham arm
  Arms: Instillation of Normal Saline

SUMMARY:
To determine if instillation of tissue plasminogen activator into a percutaneously drained intra-abdominal abscess cavity results in faster resolution of the abscess compared to normal standard of care.

DETAILED DESCRIPTION:
On day 0 Subjects will have Tissue Plasminogen Activator injected into a drainage tube and allowed to dwell in the intra-abdominal abscess for one hour before allowing it to drain by gravity. This will be repeated on day 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Intrabdominal abscess

Exclusion Criteria:

* Hypersensitivity to tPA
* Recent stroke
* Uncontrolled htn
* Recent major hemorrhage
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-07; Primary Completion 2012-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
time to eating
time to discharge
radiological evidence of resolution

SECONDARY OUTCOMES:
cost comparison

CONTACTS AND LOCATIONS:
Overall Officials: Dheeraj Rajan, MD, Principal Investigator — University Health Network - University of Toronto; Murray Asch, MD, Principal Investigator — Lakeridge Health Science Center
Locations (1):
- University Health Network, Toronto, Ontario, Canada